# **Informed Consent Form**

An Open-Label Phase 2 Trial of Acalabrutinib plus Obinutuzumab in Patients with Untreated, Low Tumor Burden Follicular Lymphoma and Other Indolent Non-Hodgkin Lymphomas

NCT Number: NCT04883437

Document IRB Approval Date: 7/22/25





# You Are Being Asked to Be in a Research Study

Concise presentation of key concepts

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study you will be one of 49 patients who are being studied, at Emory.

# Why is this study being done?

This study is being done to determine if combining two study drug therapy (called acalabrutinib and obinutuzumab) is safe and effective against your condition. You are being asked to be in this research study because you have one of the types of non-Hodgkin lymphoma that is being studied in this trial.

# Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care for your condition. Before you make your decision, you should take time to learn about the study.

# What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will participate until your disease gets worse, or the side effects of the study drugs become unacceptable, or your doctor believes the study is not in your best interest anymore, or you withdraw consent for any reason. In addition, some patients may complete the study treatment and stop taking the medications. The researchers will ask you to do the following: you will have to sign and date this informed consent form, go over your current condition, your medical history and any medications you may be taking; undergo physical examination, blood samples drawn, possible tumor biopsy, bone marrow biopsy and aspirate, imaging scans (PET/CT). You will also be requested to complete questionnaires and you will undergo a pregnancy test if you are a woman of childbearing potential. If you will participate in this research study you will receive a combination of two study treatment drugs, called: acalabrutinib and obinutuzumab. Some of these procedures will be paid for by the study.

# How is this study going to help you?

PI: Jonathon B. Cohen, MD, MS Protocol #: Winship5186-20 Page 1 of 18

Version Date: 11/14/2022 IRB Form 06162020



If you are in the study, you will be helping the researchers answer the study question. Given this is an investigational treatment, there is no guarantee that you will derive benefit if you choose to participate in this study.

# What are the risks or discomforts I should know about before making a decision?

The study will take time. The drugs that are being tested may not work any better than regular care, and may even cause harm. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious – for this study, these include: headache, muscle and joint pain, upper respiratory tract infection, bruising, infusion-related reactions, low white blood cell count, cough, constipation, diarrhea, loss of privacy, and breach of confidentiality. A full list of expected risks, their frequency and severity are in the "What are the possible risks and discomforts?" section of this document.

# Alternatives to Joining This Study

If you decide not to enter this study, there is care available to you outside of this research study. Your doctor will discuss alternative options with you. You do not have to be in this study to be treated for your cancer. Instead of being in this study, you have these options:

- 1. Treatment with other drugs, not on study
- 2. Other experimental therapies
- 3. Not doing any treatment for your lymphoma right now

#### Costs

You WILL have to pay for some of the study procedures, in particular those that are not covered by your medical insurance. In addition, the cost of the obinutuzumab (intravenous medication) will be billed to your insurance.

The study team can help you work out how much you might have to pay. There is more information in the cost section below.

# What Should I Do Next?

Read this form, or have it read to you. Make sure the study doctor or study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.) Make sure you understand which parts are research and which are standard care that you would have even if you did not join the study. Take time to consider this, and talk about it with your family and friends.



# Emory University and Saint Joseph's Hospital Consent to be a Research Subject / HIPAA Authorization

<u>Title:</u> A Multicenter, Open-Label Phase 2 Trial of Acalabrutinib plus Obinutuzumab in Patients with Untreated, Low Tumor Burden Follicular Lymphoma and Other Indolent Non-Hodgkin Lymphomas

IRB #: STUDY00002247

Principal Investigator: Jonathon B. Cohen, MD, MS

Study-Supporter: Astra Zeneca

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- · Please carefully read this form or have it read to you
- · Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### What is the purpose of this study?

You have been invited to participate in this research study because you have a form of non-Hodgkin lymphoma that is being studied in this clinical trial. This study will help study doctors find out if combining two treatments (administration of two drugs called Acalabrutinib and Obinutuzumab) is a better way to treat your cancer. The study doctors hope to learn whether the combination will be safe and will benefit you.

The two different treatments are thought to work by inhibiting two different possible ways in which a cancer cell can grow and spread:

**Obinutuzumab** has been approved by health authorities, such as the U.S. Food and Drug Administration (FDA) for the treatment or certain forms of leukemia and lymphoma. This drug is a type of antibody therapy that targets and attaches to the CD20 proteins found on lymphoma cells as well as some healthy blood cells. In people with lymphoma, CD20 may be found in higher than normal amounts.

Once attached to the CD20 protein, Obinutuzumab is thought to work in different ways, including:

- · By helping your own immune system destroy the cancer cells
- By destroying the cancer cells directly

Obinutuzumab can also harm some of your healthy immune cells that express the CD20 protein. This can put you at increased risk for infection.

**Acalabrutinib** is the name of the other drug used in this study. It's approved by the FDA for some form of Leukemia and lymphoma, but it has not been approved yet for your condition and it's currently being tested for the treatment of follicular lymphoma and other forms of non-Hodgkin lymphoma. Acalabrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals B-cells (your cancer cells) to multiply. This helps stop the spread of your cancer cells.

# What will I be asked to do?

There are three periods of the study: Screening, Study Treatment (called Induction Phase), and Follow-up.

#### Screening Period

Once you understand what is involved with participating in this study, all your questions have been answered, and you agree to take part in this research study, you will be asked to sign and date this consent form. At that point, the study doctor and the study team will look through your medical chart, ask you questions, and begin to schedule study tests and procedures. These tests and procedures will help to determine if you are eligible to take part in this study. This is called the "Screening Period".

The Screening Period of the study can take several weeks to complete. This period may include other study visits for various procedures.

The following tests and procedures will be performed by the study staff to determine if you qualify to participate in this study:

- Review of your medical history
- Review of <u>medications</u> you are currently taking and have taken in the past including herbal medications.
- A <u>physical examination</u> including measurement of your height, weight, and vital signs (temperature, respiratory rate, blood pressure, and heart rate).
- You will be asked about how well you are able to perform the normal activities of daily living; this procedure is also called assessment of <u>performance status</u>. You will be asked to answer questions about your quality of life using standard scales.
- Collection of your blood for <u>laboratory tests</u> which measure your blood chemistry (including kidney, pancreas, and liver function), count your red and white blood cells and platelets. Blood samples will also be screened for hepatitis virus testing (to test for certain viruses including those that can cause inflammation or serious infection of the liver.
- We will perform a <u>pregnancy test</u> if you are a woman who could have children. You must not be pregnant, breastfeeding, or planning to have children (male patients included) in order to join the study.



- If you have <u>tumor tissue</u> that was already taken prior to taking part in this study (archival tumor tissue), study investigator will ask for a sample of this tissue for research use and its report to be sent, if available. If archival tumor tissue is not available, you will be asked to provide fresh tumor biopsy during screening. Your study doctor can provide more information on the method that will be used to collect tumor tissue.
- Bone marrow biopsy and aspiration will be completed (if required) to help determine the status
  of your condition. This is a test where a needle is inserted into the center of the bone to collect
  a solid and liquid sample of the bone marrow
- <u>Radiographic imaging</u> by computed tomography (CT) scan or (PET/MRI) of the chest, abdomen, pelvis, and any known areas of disease will be conducted within 28 days prior to receiving treatment. These are special procedures which use X rays (CT) or magnetic resonance imaging (MRI) to create pictures of the inside of your body. These pictures will allow your study doctor to monitor your disease before, during, and after you receive study treatment.

## **Study Treatment Period**

If you qualify to participate in the study based on the results of the screening visit tests and procedures, you will be asked to return to the study doctor's office for study treatment.

If you experience any changes in your body or develop any new or worsening side effects during or after treatment, you should inform the study doctor or nurse immediately.

The following tests and procedures will be performed during treatment visits.

- You will be asked what <u>medications</u> you took or are currently taking including herbal supplements and over-the-counter medicines.
- You will be asked what <u>side-effects</u> you have experienced. You should report the
  development of any new (since your last visit) or worsening medical problems to the study
  doctor or other study staff taking care of you.
- A brief <u>physical examination</u>, including measurement of your weight.
- Your **performance status**: how well you are able to perform the normal activities of daily living
- <u>Vital signs</u> (temperature, breathing rate, blood pressure, heart rate and blood oxygen level):
- Collection of your blood for <u>laboratory tests</u> which measure your blood chemistry, including kidney and liver function, count your red and white blood cells and platelets.
- <u>Radiographic imaging</u> by computed tomography (CT) scan or magnetic resonance imaging (MRI or PET) of the chest, abdomen, pelvis, and any known areas of disease.
- You will need to undergo <u>bone marrow biopsy and aspirate</u> if required.
- You will be asked questions to assess your symptoms, and to complete <u>questionnaires</u> about your quality of life/your symptoms.
- <u>Study drugs administration</u>: Treatment will begin on Day 1 of Cycle 1. Every 28 days of the study is considered a "Cycle".

As shown in the table below, for cycles 1 and 2, you will receive acalabrutinib alone at the standard dose of 100mg orally twice daily.

For cycles 3-8, you will receive combination therapy with acalabrutinib and obinutuzumab. Obinutuzumab will be given on days 1, 8, and 15 of cycle 3 then on day 1 of cycles 4-8 (6 total cycles of obinutuzumab).

After completing treatment with obinutuzumab, you will continue on acalabrutinib alone for cycles 9 through 12.

| Treatment Cycle | Cycles 1-2 | | Cycle 3 | | | Cycle 4-8 | Cycle 9-12 |
|---|---|---|---|---|---|---|---|
| Day | 1 | 15 | 1 | 8 | 15 | 1 | 1 |
| Acalabrutinib (pill by mouth) | X | X | x | X | X | x | x |
| Obinutuzumab (by IV line) | | | X | X | X | X | |

#### Acalabrutinib

Acalabrutinib comes as a tablet to take by mouth (100mg each tablet). You will take the tablet every 12 hours (twice a day) for as long as your doctor recommends that you receive treatment. Whenever possible, take acalabrutinib at around the same times every day. Follow the directions on your prescription label carefully, and ask your doctor to explain any part you do not understand.

Swallow the tablets whole with a glass of water; do not open, chew, or break them. Acalabrutinib can be taken with or without food.

If you missed a dose, take the missed dose as soon as you remember it. However, if more than three hours have already passed since the missed dose, skip the missed dose and continue your regular dosing schedule. Do not take a double dose to make up for a missed one.

You should record on a pill diary (or patient journal) the time and date of each dose, and missed doses of acalabrutinib

Your doctor may temporarily or permanently stop your treatment or decrease your dose of acalabrutinib depending on the side effects that you experience. Be sure to talk to your doctor about how you are feeling during your treatment. Do not stop taking acalabrutinib without talking to your doctor.

#### Obinutuzumab

Each dose of obinutuzumab is 1000mg. You will receive this drug by IV line (inside the vein). If you are deemed to be at high risk for infusion-related reactions, you *may* receive the first dose of obinutuzumab as a split dose (100mg on day 1, 900 mg on day 2). This option is only available for the first dose of obinutuzumab. In this case, we would recommend that you receive the day 1 dose at 25 mg/hr x 4 hours.

## Follow-up

After completing cycle 12, you will enter the follow-up phase:

- If you had a <u>total response</u> to treatment (called CR: complete response) after cycle 12, you will be randomized (like tossing a coin) to either stop acalabrutinib treatment or to continue acalabrutinib alone until your disease gets worse, or the side effects of the study drugs become unacceptable.



- If you had a <u>partial response</u> (called PR) or your disease is stable (SD), following cycle 12, you
  will continue with acalabrutinib alone until your disease gets worse, or the side effects of the
  study drugs become unacceptable
- If your disease got <u>worse (called progressive disease PD)</u> following cycle 12, you will discontinue study treatment.

You may choose to stop any of your study drugs at any time, for any reason. When you stop or complete the study, you will have an <u>End of Study Treatment Visit</u> within 7 days of deciding to stop study treatment, a safety follow-up visit will occur after 4 weeks and then every 12 weeks for 1 year. The following tests and procedures will be performed during the follow-up visits:

- <u>Vital signs</u> (temperature, breathing rate, blood pressure, heart rate and blood oxygen level):
- A <u>physical examination</u>, including measurement of your weight
- Blood will be drawn for <u>laboratory tests</u> which measure your blood chemistry, including kidney and liver function, count your red and white blood cells and platelets.
- You will be asked what <u>medications</u> you took or are currently taking including herbal supplements and over-the-counter medicines.
- You will be asked what <u>side-effects</u> you have experienced. You should report the
  development of any new (since your last visit) or worsening medical problems to the study
  doctor or other study personnel taking care of you.
- Your <u>performance status</u>: how well you are able to perform the normal activities of daily living.
- <u>Radiographic imaging</u> by computed tomography (CT) scan or magnetic resonance imaging (MRI or PET) of the chest, abdomen, pelvis, and any known areas of disease.
- You will be asked questions to assess your symptoms, and to complete <u>questionnaires</u> about your quality of life/your symptoms.

#### How will my medicine be provided?

The medicine that you will take will be dispensed by the pharmacy and delivered to the principal investigator or study team member. The principal investigator or health care providers on his/her research team will provide the medicine to you. If you have questions about the medicine, you should ask the study doctor or study nurse. You may also call the pharmacy at if you have questions about the medicine. The number for the pharmacy is included on your medicine package.

#### Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may be still be used for this study.

#### What are the possible risks and discomforts?

There may be side effects from the study drug or procedures that are not known at this time.

#### Acalabrutinib

Acalabrutinib may cause serious side effects, including:

 Serious infections can happen during treatment with Acalabrutinib and may lead to death. Your healthcare provider may prescribe certain medicines if you have an increased risk of getting



infections. Tell your healthcare provider right away if you have any signs or symptoms of an infection, including fever, chills, or flu-like symptoms. Serious infections occur in around 10-20% of patients treated with acalabrutinib.

- Bleeding problems (hemorrhage) can happen during treatment with Acalabrutinib and can be serious and may lead to death. Your risk of bleeding may increase if you are also taking a blood thinner medicine. Tell your healthcare provider if you have any signs or symptoms of bleeding, including blood in your stools or black stools (looks like tar), pink or brown urine, unexpected bleeding or bleeding that is severe or you cannot control, vomit blood or vomit that looks like coffee grounds, cough up blood or blood clots, dizziness, weakness, confusion, changes in your speech, headache that lasts a long time, or bruising or red or purple skin marks. Minor bleeding or bruising can occur about 15% of patients treated with acalabrutinib. More serious bleeding events are rare and occur in about 1% of patients.
- Decrease in blood cell counts. Decreased blood counts (white blood cells, platelets, and red blood cells) are common with Acalabrutinib, but can also be severe. Your healthcare provider should do blood tests to check your blood counts regularly during treatment with Acalabrutinib. A low white blood cell count occurs in about 10% of patients treated with acalabrutinib.
- Second primary cancers. New cancers have happened in people during treatment with Acalabrutinib, including cancers of the skin or other organs. Your healthcare provider will check you for skin cancers during treatment with Acalabrutinib. Use sun protection when you are outside in sunlight. Secondary cancers have been observed in 5-10% of patients treated with acalabrutinib.
- Heart rhythm problems (atrial fibrillation and atrial flutter) have happened in people treated with Acalabrutinib. Tell your healthcare provider if you have any of the following signs or symptoms: fast or irregular heartbeat, dizziness, feeling faint, chest discomfort, or shortness of breath. Atrial fibrillation occurs in about 1% or less of patients treated with acalabrutinib.

The most common side effects of Acalabrutinib include headache (30%), diarrhea (30%), muscle and joint pain (20%), upper respiratory tract infection (20%), and bruising (15%).

# Side Effects Potentially Associated with Acalabrutinib

Liver Toxicity: Increases in the blood level of liver enzymes (enzymes are proteins that participate in chemical reactions in the body) may occur with acalabrutinib treatment. The role of acalabrutinib in causing the increases in these enzymes has not been established. Temporary, rarely severe liver enzyme increases have been observed in some patients treated with acalabrutinib, and these increases usually resolve with or without acalabrutinib discontinuation. Uncommonly, very high increases may potentially be associated with liver damage. You may get an increase of aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels, two major types of liver enzymes, in a blood test but not have any symptoms or feel unwell. Your study doctor will monitor your liver enzymes regularly during treatment.

#### Obinutuzumab

OBINUTUZUMAB can cause side effects that can become serious or life-threatening, including:

 Hepatitis B Virus (HBV): Hepatitis B can cause liver failure and death. If you have a history of hepatitis B infection, OBINUTUZUMAB could cause it to return. You should not receive OBINUTUZUMAB if you have active hepatitis B liver disease. Your doctor or healthcare team will screen you for hepatitis B before, and monitor you during and after, your treatment with



- OBINUTUZUMAB. Sometimes this will require treatment for hepatitis B. Symptoms of hepatitis include: worsening of fatigue and yellow discoloration of skin or eyes.
- Progressive Multifocal Leukoencephalopathy (PML): PML is a rare and serious brain infection
  caused by a virus. PML can be fatal. Your weakened immune system could put you at risk.
  Your doctor will watch for symptoms. Symptoms of PML include: confusion, difficulty talking or
  walking, dizziness or loss of balance, and vision problems. PML is very rare, occurring in less
  than 1% of patients treated with obinutuzumab.

OBINUTUZUMAB can cause side effects that may become severe or life-threatening, including:

- Infusion-Related Reactions (IRRs): These side effects may occur during or within 24 hours of any OBINUTUZUMAB infusion. Some IRRs can be serious, including, but not limited to, severe allergic reactions (anaphylaxis), acute life-threatening breathing problems, or other life-threatening IRRs. If you have a reaction, the infusion is either slowed or stopped until your symptoms are resolved. Most patients are able to complete infusions and receive medication again. However, if the IRR is life-threatening, the infusion of OBINUTUZUMAB will be permanently stopped. Your healthcare team will take steps to help lessen any side effects you may have to the infusion process. You may be given medicines to take before each OBINUTUZUMAB treatment. Symptoms of IRRs may include: fast heartbeat, tiredness, dizziness, headache, redness of the face, nausea, chills, fever, vomiting, diarrhea, rash, high blood pressure, low blood pressure, difficulty breathing, and chest discomfort. Severe infusion reactions occur in up to 10% of patients treated with OBINUTUZUMAB.
- Hypersensitivity Reactions Including Serum Sickness: Some people receiving
   OBINUTUZUMAB may have severe or life-threatening allergic reactions. This reaction may be
   severe, may happen during or after an infusion, and may affect many areas of the body. If an
   allergic reaction occurs, your doctor will stop the infusion and permanently discontinue
   OBINUTUZUMAB. Hypersensitivity reactions and serum sickness are rare.
- Tumor Lysis Syndrome (TLS): Tumor lysis syndrome, including fatal cases, has been reported in patients receiving OBINUTUZUMAB. OBINUTUZUMAB works to break down cancer cells quickly. As cancer cells break apart, their contents are released into the blood. These contents may cause damage to organs and the heart and may lead to kidney failure requiring the need for dialysis treatment. Your doctor may prescribe medication to help prevent TLS. Your doctor will also conduct regular blood tests to check for TLS. Symptoms of TLS may include nausea, vomiting, diarrhea, and tiredness. TLS is rare in patients being treated for indolent lymphomas, occurring in 1% of patients or less.
- Infections: While you're taking OBINUTUZUMAB, you may develop infections. Some of these infections may be fatal and severe, so be sure to talk to your doctor if you think you have an infection. Patients administered OBINUTUZUMAB in combination with chemotherapy, followed by OBINUTUZUMAB alone are at a high risk of infections during and after treatment. Patients with a history of recurring or chronic infections may be at an increased risk of infection. Patients with an active infection should not be treated with OBINUTUZUMAB. Serious infections occur in about 10% of patients treated with OBINUTUZUMAB.
- Low White Blood Cell Count: When you have an abnormally low count of infection-fighting
  white blood cells, it is called neutropenia. While you are taking OBINUTUZUMAB, your doctor
  will do blood work to check your white blood cell count. Severe and life-threatening
  neutropenia can develop during or after treatment with OBINUTUZUMAB. Some cases of
  neutropenia can last for more than one month. If your white blood cell count is low, your doctor
  may prescribe medication to help prevent infections. A low white blood cell count occurs in
  about 30% of patients treated with OBINUTUZUMAB.



Low Platelet Count: Platelets help stop bleeding or blood loss. OBINUTUZUMAB may reduce
the number of platelets you have in your blood; having low platelet count is called
thrombocytopenia. This may affect the clotting process. While you are taking
OBINUTUZUMAB, your doctor will do blood work to check your platelet count. Severe and lifethreatening thrombocytopenia can develop during treatment with OBINUTUZUMAB. Fatal
bleeding events have occurred in patients treated with OBINUTUZUMAB. If your platelet count
gets too low, your treatment may be delayed or reduced. Low platelet count occurs in about
10-15% of patients treated with OBINUTUZUMAB.

The most common side effects seen with Obinutuzumab in a study that included previously untreated FL patients were:

- infusion-related reactions of any severity (60%),
- low white blood cell count (10%),
- upper respiratory tract infections (50%),
- cough (30%),
- constipation (30%)
- diarrhea (30%)

# What effects could the tests have on me?

You may feel discomfort during some of these tests or may experience some inconvenience. Some may also have risks, which may include:

**Blood samples:** drawing blood from your arm may cause pain, bruising, lightheadedness, and rarely infection.

**IV line (inside the vein):** may cause discomfort, irritation, mild bruising, bleeding, leakage of drug solution, and rarely infection, nausea, and lightheadedness.

Contrast Agent Risks: Your CT or MRI procedure will require the use of a "contrast agent." The contrast agent is a substance that helps the radiologist interpret the images. The contrast agent will be injected by either a hand-held needle or a machine that does the injection. Most contrast agents stay in your body for only a few minutes, but some of them can remain for a few hours or days without any harm to you or anyone near you. Contrast agents are generally quite safe, but any injection involves some risks. The injection could harm a nerve, artery or vein, or cause infection. The contrast agent could affect kidney function or cause an allergic reaction, though these outcomes are rare. The contrast agent could also leak from your veins a little causing swelling and discomfort, that is typically treated with ice packs.

**Magnetic resonance imaging (MRI) Risks:** MRI exams use powerful magnets to create images of the body. In addition to the possible reactions to contrast materials, you may feel claustrophobic while in the magnet, and will hear loud beeping or hammering noises. If you have tattoos or any metal items in your body such as implants, pacemakers, clips or shrapnel, we will do special screening to make sure your MRI scan is done safely.

**PET/CT Risks:** For your PET/CT scan, a small amount of radioactive material will be injected by either a hand-held needle or a machine. Such injections are generally quite safe, but any injection involves some risks. The injection could harm a nerve, artery or vein, or cause infection. The radioactive material could also leak from your veins a little, causing swelling and discomfort. After



injection and a waiting period for the drug to circulate within your body, you will be asked to lie very still for several minutes while the scan takes place.

Radiation-Related Risks: You will be exposed to radiation from nuclear medicine and CT scans. These procedures are necessary for your medical care and will occur even if you do not participate in this study. The radiation dose estimate that you will receive is equal to or less than the radiation exposure allowed to be received by a radiation worker for 8 years. The principal risk associated with a radiation dose is the possibility of developing a radiation-induced cancer later in life. Although the risk from radiation is cumulative it is not expected to adversely affect your condition or treatment. The Emory University Radiation Safety Committee has reviewed and approved the use of radiation in this research study.

**Risks of biopsies:** Common side effects of a biopsy are a small amount of bleeding at the time of the procedure and mild pain in the area that was biopsied. There is also a risk for damage to structures like nerves, arteries, and veins that are near the area that is being biopsied. Infections can rarely occur after a biopsy.

If you are a woman: to protect against possible side effects of the study drug, women who are pregnant or nursing a child may not take part in this study. If you become pregnant, there may be risks to you, the embryo, or fetus. These risks are not yet known. If you are a woman of childbearing ability, you and the study doctor must agree on a method of birth control to use throughout the study and for at least 2 days after the last dose of acalabrutinib or 18 months after the last dose of obinutuzumab, whichever is longer. If you think that you have gotten pregnant during the study, you must tell the study doctor immediately. Pregnant women will be taken out of the study.

If you are a man: the effect of the study drug on sperm is not known. To protect against possible side effects, if you are a man you should not get a sexual partner pregnant while taking the study drug and for at least 2 days after the last dose of acalabrutinib or 18 months after the last dose of obinutuzumab, whichever is longer. You and the study doctor should agree on a method of birth control to use throughout the study.

Because you will be taking the study drug home, keep it out of the reach of children or anyone else who may not be able to read or understand the label. Do not let anyone else take the study drug besides you.

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

#### Will I benefit directly from the study?

This study is not designed to benefit you directly. Your condition may improve while you are in this study but it may not, and it may even get worse. This study is designed to learn more about Follicular lymphoma and other indolent Non-Hodgkin Lymphomas. The study results may be used to help others in the future.

#### Will I be compensated for my time and effort?

You will not be offered compensation for being in this study.



## What are my other options?

If you decide not to enter this study, there is care available to you outside of this research study. The study doctor will discuss these with you. You do not have to be in this study to be treated for your condition.

Taking part in this study, however, may make you unable to participate in some other research studies, if they exclude people who have taken certain treatments. You should discuss this with the researchers if you have concerns. You may wish to research other study options at websites like clinicaltrials.gov and ResearchMatch.org.

# How is my Genetic Information Protected? What are the Risks?

The Genetic Information Nondiscrimination Act (GINA) is a federal law that generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that GINA does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance, and does not apply to employers with less than 15 employees.

In addition to GINA, the State of Georgia has laws that prohibit insurers from using genetic testing information for any non-treatment purpose. However, like GINA, this state law protection has exclusions: life insurance policies, disability income policies, accidental death or dismemberment policies, Medicare supplement policies, long-term care insurance policies, credit insurance policies, specified disease policies, hospital indemnity policies, blanket accident and sickness policies, franchise policies issued on an insurance policy written as a part of workers' compensation equivalent coverage, or other similar limited accident and sickness policies.

#### Privilege

In the State of Georgia, in some circumstances your genetic information has may have special legal protections called "privilege." This means that the information cannot be used as evidence in a court. By allowing us to use and disclose your genetic information for this research study along with other information about you that genetic information used in the research may no longer have that legal protection. Other protections described in this form will still apply. There are also other confidentiality protections for research data in general under Georgia state law.

## How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.



Study records can be opened by court order. They also may be provided in response to a subpoena or a request for the production of documents.

# Storing and Sharing your Information

De-identified data from this study (data that has been stripped of all information that can identify you), including your de-identified genetic information, may be placed into public databases where, in addition to having no direct identifiers, researchers will need to sign data use agreements before accessing the data. We will remove or code any personal information that could identify you before your information is shared. This will ensure that, by current scientific standards and known methods, it is extremely unlikely that anyone would be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

Your data and specimens from this study may be useful for other research being done by investigators at Emory or elsewhere. To help further science, we may provide your deidentified data and/or specimens to other researchers. If we do, we will not include any information that could identify you. If your data or specimens are labeled with your study ID, we will not allow the other investigators to link that ID to your identifiable information.

We will use your sample and data only for research. We will not sell them. However, the results of this research might someday lead to the development of products (such as a commercial cell line, a medical or genetic test, a drug, or other commercial product) that could be sold by a company. You will not receive money from the sale of any such product.

In general, we will not give you any individual results from the study of the samples you give us. If we find something of urgent medical importance to you, we will inform you, although we expect that this will be a very rare occurrence.

# **Medical Record**

If you have been an Emory Healthcare and/or Saint Joseph's Hospital patient before, then you already have an Emory Healthcare and/or Saint Joseph's Hospital medical record. If you have never been an Emory Healthcare and/or Saint Joseph's Hospital patient, you do not have one. An Emory Healthcare and/or Saint Joseph's Hospital medical record will be made for you if an Emory Healthcare and/or Saint Joseph's Hospital provider or facility gives you any services or procedures for this study.

Copies of the consent form/HIPAA authorization that you sign will be put in any Emory Healthcare and/or Saint Joseph's Hospital medical record you have now or any time during the study.

Emory Healthcare and/or Saint Joseph's Hospital may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your Emory Healthcare and/or Saint Joseph's Hospital medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure.

The results of some study tests and procedures will be used only for research purposes and will *not* be placed in your medical record. For this study, those items include: your responses to questionnaires as well as your responses to questions about your side effects that you complete in between visits (PRO-CTCAE).

PI: Jonathon B. Cohen, MD, MS Protocol #: Winship5186-20 Page 13 of 18

Version Date: 11/14/2022 IRB Form 06162020



Tests and procedures done at non-Emory Healthcare and/or Saint Joseph's Hospital places may not become part of your Emory Healthcare and/or Saint Joseph's Hospital medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.

# In Case of Injury

If you believe you have become ill or injured from this research, you should contact Dr. Cohen at telephone number You should also let any health care provider who treats you know that you are in a research study.

If you get ill or injured from being in the study, Emory will help you to get medical treatment. Neither Emory nor the sponsor have set aside money to pay for this medical treatment. Your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurance does not pay, then you will have to pay these costs.

For Emory, the only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory employee. "Negligence" is the failure to follow a standard duty of care. You do not give up any legal rights you may have by being in this study, including any right to bring a claim for negligence.

#### Costs

The study sponsor will pay for certain items and services that you may receive if you take part in this study.

You will have to pay for the items or services for which the study sponsor does not pay. The sponsor will not pay for your regular medical care. If you have insurance, Emory Healthcare and/or Saint Joseph's Hospital will submit claims to your insurance for items and services that the sponsor does not cover. Emory will send in only those claims for items and services that it reasonably believes your insurance will pay and that the sponsor has not paid.

The actual amount that you have to pay depends on whether or not you have health insurance and whether or not that insurance will pay for any research study costs. Generally, insurance companies will not pay for items and services that are required just for a research study. Some insurance companies will not pay for regular medical treatment or treatment for complications if you are in a study. How much you will have to pay for any co-payments, deductibles or co-insurance depends on your plan. Emory and the sponsor will not pay for these costs.

It is a good idea to contact your insurance provider and tell them you want to be in this research study. Ask them what they will pay for and what they will not pay for. You can also ask the study team for help in figuring out what you will have to pay.

If you do not have insurance, Emory will review your case as part of its program for low-income patient care. The standard policies of that program will apply. The program will figure out if you have to pay any costs for taking part in the study and what those costs will be.

The study supporter (AstraZeneca) will provide acalabrutinib at no cost to the study participant. The study participant will be responsible for covering the cost of obinutuzumab.



# Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, however, you should consider the study doctor's advice about how to go off the study treatment.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

#### Authorization to Use and Disclose Protected Health Information

The privacy of your health information is important to us. We call your health information that identifies you, your "protected health information" or "PHI." To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act and regulations (HIPAA). We refer to all of these laws as the "Privacy Rules." Here we let you know how we will use and disclose your PHI for the study in which you may choose to participate.

#### PHI that Will be Used/Disclosed:

The PHI that we will use or share for the main research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.

# Purposes for Which Your PHI Will be Used/Disclosed:

We will use and share your PHI for the conduct and oversight of the research study. We will use and share your PHI to provide you with study related treatment and for payment for such treatment. We will also use and share your PHI to conduct normal business operations. We may share your PHI with other people and places that help us conduct or carry out the study, such as laboratories, data management centers, data monitors, contract research organizations, Institutional Review Boards (IRBs) and other study sites. If you leave the study, we may use your PHI to determine your health, vital status or contact information.

## Use and Disclosure of Your Information That is Required by Law:

We will use and disclose your PHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your PHI. These include subpoenas or court orders.

# Authorization to Use PHI is Required to Participate:

By signing this form, you give us permission to use and share your PHI as described in this document. You do not have to sign this form. If you do not sign this form, you may still receive non-research related treatment.

#### People Who will Use/Disclose Your PHI:

The following people and groups will use and disclose your PHI in connection with the research study:

PI: Jonathon B. Cohen, MD, MS Protocol #: Winship5186-20



- The Principal Investigator and the research staff will use and disclose your PHI to conduct the study and give you study related treatment.
- Emory Healthcare and/or Saint Joseph's Hospital may use and disclose your PHI to get payment for study related treatment and to run normal business operations.
- The Principal Investigator and research staff will share your PHI with other people and groups to help conduct the study or to provide oversight for the study.
- Dr. Jonathon Cohen is the Sponsor of the study. The Sponsor may use and disclose your PHI to make sure the research is done correctly and to collect and analyze the results of the research. The Sponsor may disclose your PHI to other people and groups like study monitors to help conduct the study or to provide oversight for the study.
- The following people and groups will use your PHI to make sure the research is done correctly and safely:
  - Emory Healthcare and/or Saint Joseph's Hospital offices that are part of the Human Research Participant Protection Program and those that are involved in study administration and billing. These include the Emory IRB, the Emory Research and Healthcare Compliance Offices, and the Emory Office for Clinical Research.
  - Government agencies that regulate the research including: Food and Drug Administration.
  - Public health agencies.
  - Research monitors and reviewer.
  - Accreditation agencies.
  - Study-supporter: AstraZeneca
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your PHI may be shared with that new institution and their oversight offices. PHI will be shared securely and under a legal agreement to ensure it continues to be used under the terms of this consent and HIPAA authorization.

# **Expiration of Your Authorization**

Your PHI will be used until this research study ends.

# **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your information. If you want to do this, you must contact the study team at:



At that point, the researchers would not collect any more of your PHI. But they may use or disclose the information you already gave them so they can follow the law, protect your safety, or make sure that the study was done properly and the data is correct. If you revoke your authorization you will not be able to stay in the study.



# Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them. The Sponsor, and people and companies working with the Sponsor on this study are not covered by the Privacy Rules. They will only use and disclose your information as described in this Consent and Authorization.

To maintain the integrity of this research study, you generally will not have access to your PHI related to this research until the study is complete. When the study ends, and at your request, you generally will have access to your PHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. If it is necessary for your health care, your health information will be provided to your doctor.

We may remove identifying information from your PHI. Once we do this, the remaining information will not be subject to the Privacy Rules. Information without identifiers may be used or disclosed with other people or organizations for purposes besides this study.

# **Contact Information**

Contact Dr. Cohen at

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or a bad reaction to the study drug, or
- if you have guestions, or concerns about the research

Contact the Emory Institutional Review Board at

- if you have questions about your rights as a research participant.
- if you have complaints about the research or an issue you rather discuss with someone outside the research team.

You may also let the IRB know about your experience as a research participant through our Research Participant Survey at



# **Consent and Authorization**

| Please <b>print</b> your name, <b>sign</b> , and <b>date</b> below if you optional studies you initialed above. By signing this cany of your legal rights. We will give you a copy of the | u agree to be in<br>consent and aut | h this research study, and any<br>horization form, you will not give up |
|---|---|---|
| Name of Subject | | |
| Signature of Subject<br>(18 or older and able to consent) | Date | : am / pm<br>Time (please circle) |
| TO BE FILLED OUT BY | STUDY TEAM | I ONLY |
| Name of Person Conducting Informed Consent I | Discussion | |
| Signature of Person Conducting Informed | Date | : am / pm<br>Time (please circle) |

**Consent Discussion**